CLINICAL TRIAL: NCT00325000
Title: An Intensive Treatment Program of Interpersonal Psychotherapy Plus Pharmacotherapy for Severely Depressed Inpatients
Brief Title: Interpersonal Psychotherapy for Severely Depressed Inpatients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: German Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHR443/4-1; SCHR443/4-2
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2000-10

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Interpersonal Psychotherapy; Sertraline; Amitriptyline

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy
Drug: sertraline or amitriptyline

SUMMARY:
We examined the hypotheses that severely depressed inpatients treated for 5 weeks with IPT-S plus pharmacotherapy have 1) a higher reduction in depressive symptoms and 2) higher response- and remission rates compared to pharmacotherapy plus CM. For the follow-up period (12 months) we hypothesized a better symptomatic and psychosocial longterm outcome and lower rates of relapse for patients initially treated with combination therapy.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted in 124 hospitalized patients with a DSM IV diagnosis of Major Depressive Disorder comparing 5 weeks of Interpersonal Psychotherapy modified for depressed inpatients (IPT-S) plus pharmacotherapy versus medication plus intensive Clinical Management (CM). The study included a prospective, naturalistic follow-up 3- and 12 months after acute treatment in 97 of 105 treatment completers. The 17-item version of the Hamilton Rating Scale for Depression (HAMD) served as the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

Major Depression (single episode, recurrent or bipolar II) according to the Structured Clinical Interview for DSM IV (SCID)and a score of ≥ 16 on the 17-item version of the Hamilton Rating Scale for Depression (HAMD)

Exclusion Criteria:

(1) concurrent diagnosis of bipolar I disorder, primary substance abuse or dependency, mental disorder due to organic factors, and borderline or antisocial personality disorder, (2) psychotic symptoms, (3) severe cognitive impairment, (4) contraindications to the study medication, and (5) being actively suicidal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11; Study Completion 2004-08

PRIMARY OUTCOMES:
The 17-item version of the Hamilton Rating Scale for Depression (HAMD) served as the primary outcome measure

SECONDARY OUTCOMES:
Beck Depression Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Berger, MD, Study Director — University Clinic Freiburg, Dept. of Psychiatry and Psychotherapy
Locations (1):
- University Clinic Freiburg , Dept. of Psychiatry and Psychotherapy, Freiburg im Breisgau, Germany